CLINICAL TRIAL: NCT07004725
Title: A Randomized, Double-blind, Prospective Study of Niacin Sustained-release Capsules in the Treatment of Rheumatoid Arthritis Complicated With Dyslipidemia
Brief Title: Therapy of Niacin for Rheumatoid Arthritis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, He Jing, Professor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Niacin RA
Record Dates: First submitted 2024-12-15; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2024-12

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Rheumatoid Arthritis (RA); niacin
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Niacin (Experimental): The first and second stage: niacin sustained-release capsules orally for 3 months
  Interventions: Drug: niacin sustained release capsules
- Placebo (Placebo Comparator): The first stage: placebo for 3 months, the second stage: niacin sustained release capsules for 3 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: niacin sustained release capsules — The first stage: the niacin group was given niacin sustained-release capsules for 3 months, and the control group was given placebo for 3 months. The second stage: Both groups were given niacin sustained-release capsules for 3 months. Dosage of niacin sustained-release capsules and placebo: 500mg once a day for week 1-4; The dose is 1000mg once a day for 5 to 12 weeks
  Arms: Niacin
Drug: Placebo — The group was given oral placebo for 3 months in the first stage and niacin sustained-release capsules for 3 months in the second stage. Dosage of niacin sustained-release capsules and placebo: 500mg once a day for week 1-4; The dose is 1000mg once a day for 5 to 12 weeks.
  Arms: Placebo

SUMMARY:
This study is a study to evaluate the safety and efficacy of administering niacin sustained-release capsules to rheumatoid arthritis with hyperlipidemia patients. Sixty patients were randomly assigned to niacin or placebo for 12 weeks, followed by niacin for 12 weeks. Changes in disease activity score, immune cell subtypes, markers of intestinal damage, intestinal flora, and other laboratory indicators will be monitored.

DETAILED DESCRIPTION:
In this study, a randomized double-blind placebo study was conducted to treat patients with rheumatoid arthritis (RA) complicated with dyslipidemia with niacin sustained-release capsules. This study intends to include 60 patients, who are randomly divided into the control group and niacin group in a 1:1 ratio. With the basic treatment of RA unchanged, the administration plan of the two groups is as follows: divided into two stages, the first stage: the niacin group is given a niacin sustained-release capsule orally for 3 months, and the control group is given a placebo orally for 3 months. The second stage: Both groups were given niacin sustained-release capsules for 3 months.The primary endpoint was the change of immune cell subsets, which clarified the immunomodulatory effect of niacin. The secondary end point was to observe the changes in blood lipid, improvement of joint symptoms, effect on intestinal barrier, the effect on intestinal flora, and safety of taking niacin sustained-release capsules.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years of age at the time of screening, weight≥35 kg.
* Diagnosed with rheumatoid arthritis satisfying the 1987 American College of Rheumatology classification criteria or ACR/EULAR 2010 classification criteria.
* Stable treatment, including DMARDs (disease-modifying anti-rheumatic drugs) and glucocorticoids, was stable in dose for at least 4 weeks, and no biological agents were used during the first 12 weeks of enrollment.
* Dyslipidemia (5.2≤TC≤7.2mmol/L, 3.4≤LDL-c≤4.9mmol/L or 1.7≤TG≤5.1 mmol/L)
* Have given written informed consent.

Exclusion Criteria:

* a. Patients with other autoimmune diseases (such as systemic lupus erythematosus, Sjogren's syndrome, ankylosing spondylitis, etc.).
* b. Patients with uncontrolled hyperuricemia and gout.
* c. Patients who take lipid-lowering drugs such as statins or fibrates orally, cardiovascular medications (such as aspirin, nitrates, calcium channel blockers, epinephrine blockers).
* d. Patients with Stevens-Johnson syndrome, toxic epidermal necrolysis, or multiple erythema.
* e. Patients with significantly impaired bone marrow function or significant anemia, leukopenia, or thrombocytopenia, excepting those secondary to active rheumatoid arthritis.
* f. Persistent or severe infection within 3 months prior to enrollment.
* g. Uncontrolled high blood pressure, diabetes, atherosclerotic cardiovascular disease, inflammatory bowel disease, peptic ulcer and other digestive diseases, end-stage diseases, or diseases that investigators believe would put patients at risk for study participation.
* h. Clinically relevant cardiovascular, liver, neurological, endocrine, or other major systemic disease that makes the implementation of the protocol or the interpretation of the findings difficult.
* i. Severe liver and kidney function impairment (severe hypoproteinemia with serum albumin <30g/L, elevated aminotransferase more than 2 times the upper limit of normal, moderate or severe renal function impairment, such as creatinine >133 μ/L, etc.).
* j. Patients with a recent and clinically severe history of drug or alcohol abuse.
* k. Pregnant.
* l. Breastfeeding.
* m. Subjects who wish to become fathers during the study or within 24 months (or 3 months washout period) after the study;
* n. Patients with congenital or acquired severe immunodeficiency, a history of cancer or lymphoproliferative disease, or patients who have received total lymphoid radiation.
* o. Known HIV-positive status.
* p. Patients with known hepatitis B or hepatitis C positive serology and patients with hepatobiliary diseases such as chronic active liver disease.
* q. Use any biologics, such as anti-tumor necrosis factor, abaxipril, tuximab, or rituximab, within 3 months prior to the first dose.
* r. Enroll in any other clinical trial involving the off-label use of investigational drugs or devices, or enroll in any other type of medical research.
* s. Body mass index (BMI) less than 18.5kg/m2 or greater than 30 kg/m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-28 (Estimated); Primary Completion 2027-01-03 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Changes in the percentages and counts of T cell subsets assessed by flow cytometry. | Baseline, 4 weeks and 12 weeks
  Evaluating changes in the percentage of regular T cell subsets in peripheral blood before and after treatment by flow cytometry.

SECONDARY OUTCOMES:
Changes in disease Activity Score in 28 joints (DAS28) assessed by physician. | Baseline,12 weeks
  Evaluating changes in DAS28 (Disease Activity Score 28) before and after treatment. DAS28 was calculated by the number of swollen joints (SJC) and tender joints (TJC) using the 28 joints count, the erythrocyte sedimentation rate (ESR) (mm/h) or c-reactive protein (CRP) (mg/L), and patient's global assessment (PGA) of disease activity.
  Compared with the baseline, a lower DAS28 would mean an improvement in disease activity. Conversely, an increase in DAS28 indicates a deterioration in disease activity.
  The specific classification of activity levels is as follows：low activity (DAS28 < 2.6), moderate activity (2.6 ≤ DAS28 ≤ 3.2), high activity (3.2 < DAS28 ≤ 5.1), and extremely high activity (DAS28 > 5.1)
Changes in the simplified disease activity index (SDAI) assessed by physician | Baseline and 12 weeks
  Evaluating changes in SDAI before and after treatment. The SDAI is a composite score based on the tender joints of 28 joints (TJC28), tender joints of 28 joints (SJC28), patients' and physicians' global assessments of disease activity, and c-reactive protein (CRP).
  Compared with the baseline, a lower SDAI would mean an improvement in disease activity. Conversely, an increase in SDAI indicates a deterioration in disease activity.
  The specific classification of activity levels is as follows：clinical remission (SDAI≤ 3.3), low activity (3.3 < SDAI≤11), moderate activity (11 < SDAI≤ 26), and high activity (SDAI> 26)
Changes in the clinical disease activity index (CDAI) assessed by physician | Baseline and 12 weeks
  Evaluating changes in CDAI before and after treatment. The Clinical Disease Activity Index (CDAI) is a composite score based on the TJC28, SJC28, and patients'and physicians'assessments.
  Compared with the baseline, a lower CDAI would mean an improvement in disease activity. Conversely, an increase in CDAI indicates a deterioration in disease activity.
  The specific classification of activity levels is as follows: clinical remission (CDAI≤ 2.8), low activity (2.8 < CDAI≤10), moderate activity (10 < CDAI≤ 22), and high activity (CDAI> 22)
ACR 20/50/70 response rate assessed by physician | Baseline and 12 weeks
  Proportion of patients with ACR20/50/70. The assessment was based on a 20%/50%/70% or greater improvement in the number of joint tenderness or joint swelling compared to baseline and a 20%/50%/70% or greater improvement in three of the remaining five core measures, which included: Patient's overall assessment of disease activity, physician's overall assessment of disease activity, patient's assessment of arthritis pain, HAQ-DI, and acute phase reactant levels (ESR vs. CRP).

OTHER OUTCOMES:
Changes of triglyceride assessed by peripheral blood physiological parameter | Baseline, 4 weeks and 12 weeks
  Evaluating the changes in triglyceride after treatment in peripheral blood.
Changes of cholesterol assessed by peripheral blood physiological parameter | Baseline, 4 weeks and 12 weeks
  Evaluating changes in cholesterol after treatment in peripheral blood.
Changes in c-reactive protein (CRP) assessed by peripheral blood physiological parameter. | Baseline, 4 weeks and 12 weeks
  Evaluating changes in concentration of CRP (mg/L) before and after treatment in peripheral blood.
Changes in erythrocyte sedimentation rate (ESR) assessed by peripheral blood physiological parameter. | Baseline, 4 weeks and 12 weeks
  Evaluating changes in concentration of ESR (mm/h) before and after treatment in peripheral blood.
Changes in serum soluble cluster of differentiation 14 (sCD14) assessed by ELISA. | Baseline, 4 weeks and 12 weeks
  Evaluating changes in sCD14 concentration in serum before and after treatment by ELISA.
Changes in serum lipopolysaccharide-binding protein (LBP) assessed by ELISA. | Baseline, 4 weeks and 12 weeks
  Evaluating changes in LBP concentration in serum before and after treatment by ELISA.
Changes in serum intestinal fatty acid-binding protein (I-FABP) assessed by ELISA.. | Baseline, 4 weeks and 12 weeks
  Evaluating changes in I-FABP concentration in serum before and after treatment by ELISA.
Numbers of participants with treatment-related adverse events assessed by questionnaire. | 12 weeks
  Adverse effects include fever, rash, abnormal liver and kidney function, new-onset infection, and any abnormal measures associated with experimental drugs were recorded by questionnaire.
Changes in intestinal flora assessed by fecal metagenomic sequencing. | Baseline and 12 weeks
  Evaluating the changes of intestinal flora before and after treatment by fecal metagenomic sequencing.